CLINICAL TRIAL: NCT05774860
Title: A Non-interventional Functional Magnetic Resonance Imaging (fMRI) and ElectroEncephalography (EEG) Study on the Neural Bases of Social Cognitive Processing in Healthy Individuals
Brief Title: Neural Bases of Social Cognitive Processing in Healthy Individuals
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Istituto Universitario di Studi Superiori Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 2197
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: social cognitive processing; empathy; mentalizing; fMRI; ageing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All healthy participants: All healthy participants will undergo behavioral assessment and fMRI or EEG
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this single center non-interventional fMRI and EEG study is to assess the neural bases of social cognitive processing in healthy individuals, and whether/how their responsiveness is modulated by ageing. The main questions it aims to answer are:

* are there specific brain regions where individual differences in social cognitive performance reflect well-established metrics of social cogntion such as empathy and mentalizing?
* is there a relationship, at the behavioral and neural levels, between ageing-related changes in social cognitive performance and empathy/mentalizing?

Healthy participants will be recruited for:

* a behavioral assessment including multiple tests of social cognition focused on empathy and mentalizing;
* for half participants: a fMRI session to collect data concerning a) brain activity associated with action observation and social cognitive processing, b) brain structural morphometriy (grey-matter volume/density), and c) brain structural connectivity (diffusion weighted imaging)
* for half participants: a EEG session to collect data concerning brain responsiveness to social cognitive processing with higher temporal resolution than that afforded by fMRI.

Results will provide an useful baseline for investigating alterations of social cognitive processing, and of their neural bases, in pathological conditions.

DETAILED DESCRIPTION:
The translational implications of results from social cognitive neuroscience are largely based on the increasing awareness on the role played by the so-called mirror and mentalizing brain networks in understanding others' behaviors and in decoding their intentions and feelings. The evidence obtained so far on the "social brain" in healthy young individuals nowadays constitutes the baseline for detecting changes in social cognitive skills associated with physiological aging or pathological conditions. The translational implications of social neuroscience are however constrained by some crucial limitations in the existing literature, that the present study aims to address. First, most the available evidence in social neuroscience results from studies assessing brain responses to the processing of single, rather than interacting, individuals. Second, most of the available knowledge concerns brain responses associated with observing others' behavior, while it is much less clear to what extent the same, or others, areas of the "social brain" are also engaged by social-related linguistic stimuli. Finally, despite the increasing emphasis on the potentially protective role of social cognition in physiological ageing, there is only preliminary evidence on possible changes of such responses in elderly individuals. On this ground, this single center non-interventional study aims to extend the available knowledge on the neural bases of social cognitive processing in 200 healthy individuals who will undergo either fMRI or EEG in association with tasks involving either visual or linguistic social stimuli concerning single and interacting individuals. In the case of EEG, data related to changes in brain electrical activity will be recorded with 64 channels. As to MRI, a multimodal session will include data concerning a) brain activity associated with social cognitive processing, b) brain structural morphometry (grey-matter volume/density), and c) brain structural connectivity (diffusion weighted imaging). Results from (f)MRI and EEG will be additionally related to individual differences in social cognitive skills, as measured through a behavioral assessment involving key variables of social cognition such as empathy (with the Balanced Emotional Empathy Scale (BEES) and the Interpersonal reactivity Index (IRI)) and mentalizing (with the Story-Based-Empathy taks and the Yoni task). MRI data will unveil the neural bases of individual differences in social cognitive performance in terms of performance-related patterns of brain activity, structure and connectivity. EEG will complement this evidence via data characterized by higher temporal resolution, to unveil the temporal development of social cognitive processes in the brain. Results will provide an useful baseline for investigating alterations of social cognition in physiological ageing and/or pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, as determined by screening assessments and principal investigator judgment
* The participant must be able to comply with study requirements as judged by the principal investigator

Exclusion Criteria:

* Any history of alcohol and/or drug abuse, addiction or suspicion of regular consumption of drugs of abuse
* Use of any psychoactive medication, or medications known to have effect on central nervous system (CNS) or blood flow
* Any contraindications for magnetic resonance imaging (MRI) scans or any brain/head abnormalities restricting MRI eligibility

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 200 healty individuals, aged 18-60 years, sampled from the general population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain activity underlying social cognitive performance at high spatial resolution | Behavioral-study day 1
  fMRI task-related data showing regional changes of brain activity associated with performing social cognitive tasks

SECONDARY OUTCOMES:
Behavioral performance 2: social cognitive skills | Behavioral-study day 1
  Participants' social cognitive skills will be assessed in terms of performance and response time in tasks requiring to process either visual or linguistic social (vs. individual) positively- and negatively-valenced stimuli inducing variable degree of arousal.
Brain activity underlying social cognitive performance at high temporal resolution | Behavioral-study day 1
  EEG task-related data showing the temporal development of the neural processes associated with performing social cognitive tasks
Behavioral performance 1: empathy and mentalizing | Behavioral-study day 1
  Participants' disposition towards social stimuli will be assessed in terms of well-know metrics such as affective empathy or cognitive empathy (as measures with the Balanced Emotional Empathy Scale (BEES) or the Interpersonal Reactivity Index (IRI)), or mentalizing (as measured with the Story-Based Empathy task)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Ita, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Requests for sharing will assessed case by case, and data will be made available on reasonable request.